CLINICAL TRIAL: NCT01294319
Title: Evaluation of Cortisol Resistance in Young Sedentary and Endurance-trained Men and Elderly Sedentary Men
Brief Title: Evaluation of Cortisol Resistance in Young Sedentary and Endurance-Trained Men
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 110078; 11-CH-0078 (Other: National Institutes of Health)
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Results first posted 2017-11-21 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Cortisol Resistance; Negative Feedback; ACTH; Mineralcorticoid; Glucocorticoid
Keywords: Cortical Resistance; ACTH; Glucocorticoid; Mifepristone; SPIRONOLACTONE; Exercise; Hypothalamic-Pituitary-Adrenal Axis; Healthy Volunteer; HV
MeSH Terms: conditions — Motor Activity | interventions — Mifepristone; Spironolactone; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Sedentary young adults, SMCP (Experimental): Spironolactone, Then Mifepristone, Then Combined, Then Placebo (SMCP), Then Dexamethasone
  Interventions: Drug: Mifepristone; Drug: Placebo; Drug: Spironolactone; Drug: Combined; Drug: Dexamethasone
- Endurance-trained young athletes, SMCP (Experimental): Spironolactone, Then Mifepristone, Then Combined, Then Placebo (SMCP), Then Dexamethasone
  Interventions: Drug: Mifepristone; Drug: Placebo; Drug: Spironolactone; Drug: Combined; Drug: Dexamethasone
- Sedentary young adults, MSPC (Experimental): Mifepristone, Then Spironolactone, Then Placebo, Then Combined (MSPC), Then Dexamethasone
  Interventions: Drug: Mifepristone; Drug: Placebo; Drug: Spironolactone; Drug: Combined; Drug: Dexamethasone
- Endurance-trained young athletes, MSPC (Experimental): Mifepristone, Then Spironolactone, Then Placebo, Then Combined (MSPC), Then Dexamethasone
  Interventions: Drug: Mifepristone; Drug: Placebo; Drug: Spironolactone; Drug: Combined; Drug: Dexamethasone
- Sedentary young adults, CPSM (Experimental): Combined, Then Placebo, Then Spironolactone, Then Mifepristone (CPSM), Then Dexamethasone
  Interventions: Drug: Mifepristone; Drug: Placebo; Drug: Spironolactone; Drug: Combined; Drug: Dexamethasone
- Endurance-trained young athletes, CPSM (Experimental): Combined, Then Placebo, Then Spironolactone, Then Mifepristone (CPSM), Then Dexamethasone
  Interventions: Drug: Mifepristone; Drug: Placebo; Drug: Spironolactone; Drug: Combined; Drug: Dexamethasone
- Sedentary young adults,PCMS (Experimental): Placebo, Then Combined, Then Mifepristone, Then Spironolactone (PCMS), Then Dexamethasone
  Interventions: Drug: Mifepristone; Drug: Placebo; Drug: Spironolactone; Drug: Combined; Drug: Dexamethasone
- Endurance-trained young athletes,PCMS (Experimental): Placebo, Then Combined, Then Mifepristone, Then Spironolactone (PCMS), Then Dexamethasone
  Interventions: Drug: Mifepristone; Drug: Placebo; Drug: Spironolactone; Drug: Combined; Drug: Dexamethasone

INTERVENTIONS:
Drug: Mifepristone
  Other Names: Mifepristone 400 MG
Drug: Placebo
Drug: Spironolactone
  Other Names: Spironolactone 200 MG
Drug: Combined
  Other Names: Mifepristone 400 MG and Spironolactone 200 MG
Drug: Dexamethasone
  Other Names: Dexamethasone 0.25 mg

SUMMARY:
This study proposes to examine multiple aspects of the hypothalamic-pituitary-adrenal axis in younger endurance trained and sedentary men, and in older sedentary men.

DETAILED DESCRIPTION:
Adrenocorticotropin (ACTH) secretion is normally exquisitely regulated through endogenous stimulation by corticotrophin-releasing hormone (CRH) and negative feedback inhibition by cortisol, resulting in a circadian rhythm of cortisol. Recent evidence suggests that older men, and younger men who are endurance-trained athletes, both have reduced sensitivity to negative feedback, and perhaps increased basal levels of cortisol and ACTH. To investigate these possibilities, we propose to examine multiple aspects of the hypothalamic-pituitary-adrenal axis in younger endurance trained and sedentary men, and in older sedentary men.

Subjects will collect saliva during two evenings before additional testing, and will on the same evening collect urine for twelve hours, both for cortisol measurements. Blood samples will be collected to evaluate the response to dexamethasone. We also will assess ACTH and cortisol responses to medications that reduce negative inhibition of ACTH. This testing will occur in the evening and will include administration of the glucocorticoid antagonist mifepristone, the mineralocorticoid antagonist spironolactone, and/or a look-alike tablet, on four occasions.

ELIGIBILITY:
* INCLUSION CRITERIA:

Men aged 18 to 30 years of age are required for the young endurance trained and sedentary groups; men aged 65-80 years for the older study group, who will meet criteria for sedentary men below. Women and children are excluded to enhance homogeneity of responses and avoid the influence of menstrual cyclicity on the HPA axis.

Sedentary:

* Less than one hour physical activity per week for three years
* No change in exercise anticipated for 6 weeks

Trained:

* Greater than 45km (28 miles) running per week for at least 3 months
* No change in exercise anticipated for 6 weeks

For all participants:

* All races
* Sleep-wake cycle with sleeping at night, wakening between 5 and 8 AM
* BMI between 18 and 25 kg/M2
* Normal TSH and free T4

EXCLUSION CRITERIA:

For all participants:

* Sleep disorders as assessed by sleep apnea questionnaire
* Smoking
* No more than 2 servings of alcohol daily
* Medications known to affect the HPA axis or steroid metabolism, including narcotics, Glucocorticoids, megace or CYP3A4 modulators
* History of psychiatric or endocrine disorders
* Marijuana or other illicit drug use
* Recent appendicular or skeletal injury
* Uncontrolled hypertension
* Chronic pain requiring daily medication
* Current treatment with medications related to mineralocorticoid function such as potassium, ACE-inhibitors, ARBs, diuretics, spironolactone
* Frailty score of 4-7 on the Canadian Study of Health and Aging frailty scale (Rockman 2005)
* Overtraining syndrome will be an exclusion and will be assessed by questionnaire
* Abnormal creatinine level (greater than 1.2 mg/dl)
* Liver function tests greater than two fold normal
* Benzodiazepine use

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2011-01-24; Primary Completion 2016-08-10 (Actual); Study Completion 2016-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynnette K Nieman, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bauer ME. Stress, glucocorticoids and ageing of the immune system. Stress. 2005 Mar;8(1):69-83. doi: 10.1080/10253890500100240. PMID 16019599
- [Background] Bertagna X, Bertagna C, Luton JP, Husson JM, Girard F. The new steroid analog RU 486 inhibits glucocorticoid action in man. J Clin Endocrinol Metab. 1984 Jul;59(1):25-8. doi: 10.1210/jcem-59-1-25. PMID 6327758
- [Background] Booth CK, Probert B, Forbes-Ewan C, Coad RA. Australian army recruits in training display symptoms of overtraining. Mil Med. 2006 Nov;171(11):1059-64. doi: 10.7205/milmed.171.11.1059. PMID 17153542
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-CH-0078.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Sedentary Young Adults, SMCP; Endurance-trained Young Athletes, SMCP: Spironolactone, Then Mifepristone, Then Combined, Then Placebo, Then Dexamethasone
- Sedentary Young Adults, MSPC; Endurance-trained Young Athletes, MSPC: Mifepristone, Then Spironolactone, Then Placebo, Then Combined, Then Dexamethasone
- Sedentary Young Adults, CPSM; Endurance-trained Young Athletes, CPSM: Combined, Then Placebo, Then Spironolactone, Then Mifepristone, Then Dexamethasone
- Sedentary Young Adults,PCMS; Endurance-trained Young Athletes,PCMS: Placebo, Then Combined, Then Mifepristone, Then Spironolactone, Then Dexamethasone
Period: Overall Study
Arm/Group | Sedentary Young Adults, SMCP | Endurance-trained Young Athletes, SMCP | Sedentary Young Adults, MSPC | Endurance-trained Young Athletes, MSPC | Sedentary Young Adults, CPSM | Endurance-trained Young Athletes, CPSM | Sedentary Young Adults,PCMS | Endurance-trained Young Athletes,PCMS
Started | 4 | 6 | 5 | 5 | 5 | 4 | 5 | 5
Completed | 4 | 6 | 5 | 5 | 5 | 4 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sedentary Young Adults, SMCP | Endurance-trained Young Athletes, SMCP | Sedentary Young Adults, MSPC | Endurance-trained Young Athletes, MSPC | Sedentary Young Adults, CPSM | Endurance-trained Young Athletes, CPSM | Sedentary Young Adults,PCMS | Endurance-trained Young Athletes,PCMS | Total
Number analyzed (Participants) | 4 | 6 | 5 | 5 | 5 | 4 | 5 | 5 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.57 (0.99) | 25.01 (1.58) | 24.2 (2.33) | 25.2 (1.79) | 23.3 (2.97) | 24.5 (4.22) | 27.8 (3.06) | 23.6 (4.01) | 24.73 (2.87)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 4 | 5 | 5 | 5 | 4 | 4 | 5 | 5 | 37
  Unknown | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Body Mass Index [Mean (Standard Deviation); unit: Kg/m^2] | 23.6 (4.33) | 24.0 (3.27) | 23.7 (3.04) | 22.3 (1.89) | 24.2 (2.75) | 24.1 (1.10) | 23.4 (2.98) | 22.8 (2.00) | 23.53 (2.63)
Race [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 2 | 1 | 0 | 1 | 1 | 0 | 7
  Black | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 4
  White | 1 | 3 | 2 | 4 | 2 | 2 | 2 | 1 | 17
  Unknown | 2 | 2 | 1 | 0 | 1 | 0 | 1 | 4 | 11
Total Fat Percent [Mean (Standard Deviation); unit: percent] | 21.1 (6.90) | 20.2 (5.16) | 25.2 (5.11) | 19.5 (1.99) | 23.2 (5.82) | 19.7 (5.15) | 24.4 (5.16) | 16.8 (4.04) | 21.33 (5.28)
Fat mass [Mean (Standard Deviation); unit: kg] | 16.28 (8.05) | 16.73 (5.60) | 19.13 (4.80) | 14.70 (3.19) | 19.21 (8.69) | 15.13 (3.79) | 17.64 (4.31) | 13.69 (4.56) | 16.61 (5.45)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Suppressors After Dexamethasone
Description: All subjects will take 0.25mg dexamethasone as an outpatient between 2300 and 2400h and will then report to the clinic by 0800h next day for the final visit.
  At the final visit, cortisol response to dexamethasone suppression was assessed. The cortisol response was dichotomized (suppression vs. non-suppression, using 1.8 ug/dL as the cutoff point) and compared between the two groups,Sedentary Young Adults and Endurance-trained Young Athletes.
Time Frame: cortisol measured between 8 and 9 after dexamethasone was taken between 11 PM and midnight
Measure: Count of Participants; unit: Participants
Groups:
- Endurance-trained Young Athletes: Endurance-trained Young Athletes group consists of 20 subjects, each subject was randomized to one of the following four arms:
  1. Spironolactone, Then Mifepristone, Then Combined, Then Placebo, Then Dexamethasone
  2. Mifepristone, Then Spironolactone, Then Placebo, Then Combined, Then Dexamethasone
  3. Combined, Then Placebo, Then Spironolactone, Then Mifepristone, Then Dexamethasone
  4. Placebo, Then Combined, Then Mifepristone, Then Spironolactone, Then Dexamethasone
- Sedentary Young Adults: Sedentary young adults group consists of 19 subjects, each subject was randomized to one of the following four arms:
  1. Spironolactone, Then Mifepristone, Then Combined, Then Placebo, Then Dexamethasone
  2. Mifepristone, Then Spironolactone, Then Placebo, Then Combined, Then Dexamethasone
  3. Combined, Then Placebo, Then Spironolactone, Then Mifepristone, Then Dexamethasone
  4. Placebo, Then Combined, Then Mifepristone, Then Spironolactone, Then Dexamethasone
Arm/Group | Endurance-trained Young Athletes | Sedentary Young Adults
Number analyzed (Participants) | 20 | 19
Participants | 0 | 1
Statistical Analysis 1: Comparison: Endurance-trained Young Athletes vs Sedentary Young Adults; Test type: Superiority; p = 0.4872, Fisher Exact

2. Secondary Outcome: Post-dexamethasone Cortisol Level
Time Frame: Cortisol obtained at 8-9 AM after dexamethasone taken between 11 pm and midnight
Measure: Mean (Standard Deviation); unit: mcg/dL
Arm/Group | Endurance-trained Young Athletes | Sedentary Young Adults
Number analyzed (Participants) | 20 | 19
mcg/dL | 11.98 (5.92) | 9.98 (5.39)
Statistical Analysis 1: Comparison: Endurance-trained Young Athletes vs Sedentary Young Adults; Test type: Superiority; p = 0.2786, t-test, 2 sided

ADVERSE EVENTS:
Groups:
- Sedentary Young Adults: Sedentary young adults group consists of 19 subjects, each subject was randomized to one of the following four arms:
  Spironolactone, Then Mifepristone, Then Combined, Then Placebo, Then Dexamethasone Mifepristone, Then Spironolactone, Then Placebo, Then Combined, Then Dexamethasone Combined, Then Placebo, Then Spironolactone, Then Mifepristone, Then Dexamethasone Placebo, Then Combined, Then Mifepristone, Then Spironolactone, Then Dexamethasone
- Atheletes: Endurance-trained Young Athletes group consists of 20 subjects, each subject was randomized to one of the following four arms:
  Spironolactone, Then Mifepristone, Then Combined, Then Placebo, Then Dexamethasone Mifepristone, Then Spironolactone, Then Placebo, Then Combined, Then Dexamethasone Combined, Then Placebo, Then Spironolactone, Then Mifepristone, Then Dexamethasone Placebo, Then Combined, Then Mifepristone, Then Spironolactone, Then Dexamethasone
Arm/Group | Sedentary Young Adults | Atheletes
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 0/19 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No